CLINICAL TRIAL: NCT06270667
Title: The LYMfit Study: Exercise Training to Prevent Cardiovascular Disease in Lymphoma Survivors
Brief Title: Effects of Exercise Training in Survivors of Lymphoma
Acronym: LYMfit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Tormod Skogstad Nilsen, Principal Investigator, PhD, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LYMfit
Record Dates: First submitted 2024-01-19; First posted 2024-02-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma; Physical Exercise; Cardiotoxicity; Cardiovascular Diseases; Chemotherapeutic Toxicity
MeSH Terms: conditions — Lymphoma; Motor Activity; Cardiotoxicity; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Exercise (Experimental): Aerobic Exercise twice weekly for 5 months.
  Interventions: Behavioral: Aerobic Exercise
- Combined Aerobic and Resistance Exercise (Experimental): Combined Aerobic and Resistance Exercise twice weekly for 5 months.
  Interventions: Behavioral: Combined Aerobic and Resistance Exercise
- Standard Care (No Intervention): Standard Care, i.e no exercise intervention.
- Reference Aerobic Exercise (Active Comparator): Aerobic Exercise twice weekly for 5 months.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants receive twice weekly supervised aerobic treadmill-based exercise sessions for five months. Session duration varies from 20 to 60 minutes, including warm-up, with exercise intensity ranging from 60 to 95% of peak heart rate. Maximal exercise capacity (VO2peak and peak heart rate) will be determined by the CPET performed by certified exercise physiologists at baseline.The exercise prescription will be sequenced so that the exercise intensity and -duration of each exercise varies within each week, leading to an accumulative increase in weekly exercise volume throughout the intervention. This intervention is also given to the Active Comparator group (i.e. non-cancer reference group)
  Arms: Aerobic Exercise; Reference Aerobic Exercise
Behavioral: Combined Aerobic and Resistance Exercise — Twice weekly, supervised combined aerobic and resistance exercise sessions will be offered to participants. Participants randomized to the combined aerobic and resistance training group will follow the same aerobic exercise prescription as described for the Aerobic Exercise arm. In addition, participants in this group will perform five resistance exercises after the aerobic sessions. The resistance exercises will be leg press, knee extension, and calf rise, followed by seated row and chest press. Following familiarization, the training load will progressively increase following a linear periodization model throughout the intervention. exercise prescription will be sequenced so that the exercise intensity and -duration of each exercise varies within each week, leading to an accumulative increase in weekly exercise volume throughout the intervention. Only Lymphoma participants can be randomized to this arm.
  Arms: Combined Aerobic and Resistance Exercise

SUMMARY:
This study aims to compare the effects of aerobic exercise with or without addition of resistance exercise to usual care in individuals treated with anthracyclines for lymphomas and to compare exercise effects to age- and sex-matched individuals with no prior history of malignant diseases.

DETAILED DESCRIPTION:
In this study, a comparison of the exercise effects between individuals previously treated for specific lymphoma diagnoses and individuals with no history of cancer will be conducted. Therefore, in addition to a randomized controlled trial in individuals with a previous lymphoma diagnosis (i.e., exercise groups and a non-exercising control group), a reference group comprising age- and sex-matched individuals with no history of a cancer diagnosis will also be included. Participants in the reference group will undergo the same exercise intervention as the aerobic exercise group. This study recruits through invitation only.

The primary endpoint in this study is the change in cardiorespiratory fitness, assessed as VO2peak. Secondary endpoints include common risk factors for cardiovascular disease and cardiometabolic health, other variables derived from the cardiopulmonary exercise test and lung function assessments, and muscle cellular endpoints from muscle biopsies obtained from m. vastus lateralis, in addition to patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria Lymphoma participants:

* Listed in relevant registers
* Confirmed lymphoma diagnosis (i.e., Hodgkin lymphoma and aggressive non-Hodgkin lymphoma)
* Completed treatment in the past two to five years without relapse or second cancer
* Previous anthracycline treatment with or without mediastinal radiation
* No severe cancer-related fatigue (per self-report)

Inclusion Criteria Lymphoma participants and non-cancer reference group:

* Currently not performing >75 minutes/week of aerobic exercise
* Willing and able to adhere to all study procedures.

Exclusion Criteria Lymphoma participants:

* Relapse since diagnosis
* A history, or current presence, of another diagnosis of invasive cancer of any kind

Exclusion Criteria Lymphoma participants and non-cancer reference group:

* Presence of any uncontrolled- or recent cardiovascular disease
* Has undergone heart surgery
* Uses a pacemaker
* Pregnancy
* Unable to read and understand Swedish (applicable for the Swedish site only)
* Unable to read and understand Norwegian (applicable for the Norwegian site)
* Any physical or mental health condition restricting adherence to study protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
VO2peak | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Peak oxygen uptake during a treadmill-based cardiopulmonary exercise test

SECONDARY OUTCOMES:
Systolic- and diastolic heart chamber dimensions | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Cardiac morphology and function will be assessed by echocardiography (2D and 3D echocardiography and 2D strain echocardiography)
Systolic- and diastolic longitudinal strain | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Cardiac morphology and function will be assessed by echocardiography (2D and 3D echocardiography and 2D strain echocardiography)
Lean body mass | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Body composition will be assessed by dual x-ray absorptiometry
Fat mass | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Body composition will be assessed by dual x-ray absorptiometry
Forced Vital Capacity | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Lung function are assessed with spirometry.
Forced Expiratory Volume 1 sec | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Lung function are assessed with spirometry.
Maximal voluntary ventilation | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Lung function are assessed with spirometry.
Diffusion capacity | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Diffusion capacity for carbon monoxide is assessed with single breath diffusion capacity test.
Physical activity | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Actigraph accelerometer with physical activity diary. 7 days consecutive measurement at each timepoints.
Physical activity | Baseline, 10-12 weeks from baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Patient reported physical activity is assessed with Godin Leisure-Time Exercise Questionnaire
Global Health related Quality of life | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Patient reported health related quality of life will be assessed with EORTC QLQ C 30
Blood volume | Baseline, five months from baseline (i.e. end of intervention) and 2 years from baseline
  Will be assessed in Norway only. Using the carbon monoxide rebreathing method.
Muscle fiber area | Baseline, five months from baseline (i.e. end of intervention)
  Will be assessed in Norway only. Change in muscle morphology will be assessed in muscle biopsies using immunohistochemistry
Muscle fiber type | Baseline, five months from baseline (i.e. end of intervention)
  Will be assessed in Norway only. Change in muscle morphology will be assessed in muscle biopsies using immunohistochemistry
Muscle mitochondria mass | Baseline, five months from baseline (i.e. end of intervention)
  Will be assessed in Norway only. Change in mitochondrial proteins will be assessed in muscle biopsies using western blot

OTHER OUTCOMES:
Muscle genome-wide DNA methylation and gene expression | Baseline, five months from baseline (i.e. end of intervention)
  Will be assessed in Norway only. For a sub-group of participants, muscle biopsies will be further processed for RNA and DNA
Adverse events | Five months from baseline (i.e. end of intervention)
  Medical records and Patient reported outcome version of the Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Tormod S. Nilsen, PhD, Principal Investigator — Norwegian School of Sport Sciences
Locations (2):
- Norweigan School of Sport Sciences, Oslo, Norway
- Helena Igelström, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No